CLINICAL TRIAL: NCT03827226
Title: Breech External Cephalic Version Intervention Trial- A Prospective Study
Brief Title: Breech External Cephalic Version Intervention Trial
Acronym: BREXIT
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Larry Hinkson, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA2/241/18
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Breech Presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective study assessing the use of external cephalic version for the management of breech presentation in pregnancy.

DETAILED DESCRIPTION:
The primary aim of the study is to determine the success rate of external cephalic version for breech presentation from 36 gestational weeks.

ELIGIBILITY:
Inclusion Criteria:

* Presence of the written consent of the patients.
* The patients must be over 18 years old .
* No limit in the ability to consent.

Exclusion criteria:

* Age under 18
* Limited ability to consent
* Placenta previa
* Fetal abnormalities

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients presenting with breech presentation to the antenatal clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of external cephalic version | 4 hours after external cephalic version
  Mean Percentage (Range 0-100) - Successfully performed external cephalic Versions / Total number of participants,

SECONDARY OUTCOMES:
Sonographic Fetal Parameters: Head Circumference | 30 Minutes before external cephalic version
  Measurements in mm
Sonographic Fetal Parameters: Abdominal Circumference | 30 Minutes before external cephalic version
  Measurements in mm
Sonographic Fetal Parameters: Femur length | 30 Minutes before external cephalic version
  Measurements in mm
Sonographic Fetal Parameters: Amniotic Fluid | 30 Minutes before external cephalic version
  Measurements in mm
Fetal Doppler Indices middle cerebral | 30 Minutes before external cephalic version
  Index Measurements/Ratios
Fetal Doppler Indices Umbilical Pulsatility Index | 30 Minutes before external cephalic version
  Index Measurements/Ratios
Fetal Doppler Indices Umbilical Resistance Index | 30 Minutes after external cephalic version
  Index Measurements/Ratios
Maternal Doppler Indices Uterine artery Right | 30 Minutes before external cephalic version
  Index Measurements/Ratios
Maternal Doppler Indices Uterine artery Left | 30 Minutes after external cephalic version
  Index Measurements/Ratios
Bladder volume | 30 Minutes before external cephalic version
  Volume measurement
Distance Symphysis to Breech | 30 Minutes before external cephalic version
  mm
Depression and Anxiety Stress scale score | 60 minutes before external cephalic version
  A scale score with a range from 0 to 42 (0-10 is normal and 35-42 extremely severe)
Depression and Anxiety Stress scale score | 120 Minutes after external cephalic version
  A scale score with a range from 0 to 42 (0-10 is normal and 35-42 extremely severe)
Fetal reflexes | 30 Minutes before external cephalic version
  Percentage
Mode of delivery | 6 weeks after delivery
  Type of delivery Vaginal or Caesarean
Incidence of fetal extended legs | 30 Minutes before external cephalic version
  Numerical percentage
Incidence of bleeding | 30 minutes after external cephalic version
  Numerical percentage
Incidence of ruptured membranes | 30 minutes after external cephalic version
  Numerical percentage
Incidence of pathological Cardiotocogram | 30 minutes after external cephalic version
  Numerical percentage
Incidence of emergency delivery | 30 minutes after external cephalic version
  Numerical percentage
Pain scores | 30 minutes after external cephalic version
  Numerical score. Pain scale Linkert score. (0-10 with 10 being extremely painful)
Incidence of tocolysis | 30 minutes after external cephalic version
  Numerical percentage
Incidence of umbilical cord looping | 30 Minutes before external cephalic version
  Numerical percentage

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hinkson, FRCOG, Principal Investigator — Consultant in Obstetrics
Locations (1):
- Charité University Hospital, Mitte, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmeyr GJ, Kulier R. External cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2000;(2):CD000083. doi: 10.1002/14651858.CD000083. PMID 10796122
- [Result] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins--Obstetrics. Practice Bulletin No. 161: External Cephalic Version. Obstet Gynecol. 2016 Feb;127(2):e54-61. doi: 10.1097/AOG.0000000000001312. PMID 26942387
- [Result] External Cephalic Version and Reducing the Incidence of Term Breech Presentation: Green-top Guideline No. 20a. BJOG. 2017 Jun;124(7):e178-e192. doi: 10.1111/1471-0528.14466. Epub 2017 Mar 16. No abstract available. PMID 28299867
- [Derived] Schauer M, Latartara E, Alonso-Espias M, Rossetti E, Gebert P, Henrich W, Hinkson L. Depression, anxiety and stress in women with breech pregnancy compared to women with cephalic presentation-a cross-sectional study. Arch Gynecol Obstet. 2023 Feb;307(2):409-419. doi: 10.1007/s00404-022-06509-0. Epub 2022 Mar 27. PMID 35344082